CLINICAL TRIAL: NCT04683380
Title: Study of the Robustness Predictive Factors in People Aged Over 75 Years After Going to the Emergency Room
Brief Title: Robustness Predictive Factors in People Aged Over 75 Years After Going to the Emergency Room (ROB-U)
Acronym: ROB-U
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0099
Record Dates: First submitted 2020-12-16; First posted 2020-12-24 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Aging; Emergency Room; Risk Factors
Keywords: Elderly dependence; Emergency room visits; Lack of autonomy; Robustness; Re-hospitalization
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
After emergency room visits, the elderly patients can increase their dependence and functional decline. In this context the goal of this study is to demonstrate that there are robustness predictive factors after visit to the emergency room.

DETAILED DESCRIPTION:
The emergency department is one of the main access routes to the hospital for elderly patients.

Older age is often associated with an increase risk of longer stay in the emergency room with a high subsequent risk of hospital re-admission. One of the essential care objectives when treating these patients is to maintain the autonomy to avoid any dependence in order to keep the quality of life, and limit the time of hospitalization.

Emergency room visits and hospitalizations are too often considered as a source of autonomy loss aggravation in the elderly. Many studies have demonstrated the mortality predictive factors existence, functional decline, or re-hospitalization of the elderly after an emergency room visit or after hospitalization.

No study until now has investigated the existence of factors directly predictive of robustness. Then the goal of this study is to demonstrate that there are robustness predictive factors after going to the emergency room.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the emergency room
* Patients aged ≥ 75 years old
* Patients without cognitive disorders or vigilance disorders
* Patients living at home
* Patients able to give its non-opposition

Non inclusion Criteria:

* Patients admitted to the hospital in the last 3 months
* Patients refusing to participate in the study

Exclusion Criteria:

* Patients whose stay is < 14h or > 48h
* Patients who die during hospitalization
* Patient not hospitalized
* Patient not returning home after discharge from hospital

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population is composed of patients aged more than 75 years old and who have eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Identification of predictive factors of robustness : Autonomy level at home (ADL score) | 3 months
  ADL self-performance coding ranges from 0 (independent) to 4 (total dependence).
Identification of predictive factors of robustness by a questionnaire (help at home) | 3 months
  Need of help at home such as : toilet, breakfast, lunch, dinner (yes or not)
Identification of predictive factors of robustness by a questionnaire (family visits) | 3 months
  Number of family visits
Identification of predictive factors of robustness by a questionnaire (appetit) | 3 months
  loss of appetite (yes or not)
Identification of predictive factors of robustness (heart rate) | 3 months
  Heart rate during hospitalization (minimum and maximum values)
Identification of predictive factors of robustness (Modified Triage Risk Screening Tool (TRST)) score | 3 months
  The TRST score is a tool to predict repeat emergency department visits and hospitalizations in older patients discharged from the emergency department; This tool evaluates 5 dimensions : cognitive disorders presence, walking disorders, polymedication, hospitalization antecedents and functional assessment (loss of autonomy). Every dimension is worth 1 point if the patient presents the disorder. The final maximum score is 5 points.
Identification of predictive factors of robustness : BMI (Body Mass Index) | 3 months
  Body mass index
Albuminemia | 3 months
  Rate of Albuminemia
Identification of predictive factors of robustness : Lifestyle | 3 months
  Lifestyle: person living alone (yes or not)
Sleep assessment using a Visual Analog Scale (VAS). | 3 months
  This scale allows patients to assess their fatigue. The patients locate their fatigue intensity on a 100-millimeters horizontal line. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
Rate of re-hospitalization | 3 months
  Only direct re-hospitalizations in emergency rooms and geriatric short stay will be counted
Rate of patient survival | 3 months
  Rate of patient survival
Rate of lack of Institutionalization | 3 months
  Rate of lack of Institutionalization

CONTACTS AND LOCATIONS:
Overall Officials: Jean Bouquillon, Principal Investigator — Hôpital Saint-Vincent de Paul
Locations (1):
- Saint-Vincent Hospital, Lille, Haut-de-France, France

IPD SHARING:
Plan to Share IPD: No